CLINICAL TRIAL: NCT02102516
Title: A Single Arm, Open Label Study of the Safety, Efficacy, and Pharmacokinetics of SPRIX (Intranasal Ketorolac Tromethamine) in 0 to 11 Year-Old Patients Undergoing Open Surgical Procedures
Brief Title: SPRIX in 0 to 11 Year-Old Patients Undergoing Open Surgical Procedures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Egalet Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1SPR11002
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Pain
Keywords: Post operative pain management
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SPRIX(intranasal ketorolac tromethamine) (Experimental): Based on subject weight
  Interventions: Drug: SPRIX(intranasal ketorolac tromethamine)

INTERVENTIONS:
Drug: SPRIX(intranasal ketorolac tromethamine) — Dose: Subjects weighing 3.0 kg received 3.15 mg (1 spray/1 nostril), subjects weighing 5.1 - 10.0 kg received 5.25 mg (1 spray/1 nostril), subjects weighing 10.1 - 15.4 kg received 10.5 mg (1 spray/1 nostril), subjects weighing 15.5 - 31.7 kg received 15.75 mg (1 spray/1 nostril), and subjects weighing >=31.8 kg received 31.5 mg (1 spray/2 nostrils).
  Duration of Treatment: Subjects received a dose of SPRIX every 6 hours from the day of surgery until the morning of post-operative Day 2. Dosing may have resumed after final PK assessment of the morning of post-operative Day 3 until post-operative Day 4. A follow-up phone interview took place 14 days after the final dose of study drug.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics and safety of postoperative administration of SPRIX in pediatric patients (ages 0-11) undergoing open surgical procedures.

DETAILED DESCRIPTION:
Evaluate the pharmacokinetics and safety of postoperative administration of SPRIX in pediatric patients (ages 0-11) undergoing open surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients ages 0 to 11 years.
* Undergoing an open surgical procedure expected to result in at least moderate pain based on an age appropriate scale.
* Body mass index (BMI) ≤ 95th percentile of age.
* Surgical procedures that would allow the subject to likely remain in the hospital until the morning of post-operative day 3 (to complete PK sample collection).
* With parental assistance, willing and able to complete the study procedures and pain scales and to communicate meaningfully with the study personnel.
* In generally good health and capable of undergoing surgery.
* Females at risk of pregnancy were to use an acceptable form of birth control and have a negative serum or urine pregnancy test (although it is anticipated that all 0-11 year old subjects will be pre-menarchal).
* Willing to refrain from use of non-study analgesics for the duration of the study, from the day of surgery up to post-operative Day 4.
* Assents to participation and his/her parent or guardian is willing and able to sign the informed consent approved by the IRB.

Exclusion Criteria:

* Surgical procedure performed exclusively by laparoscopy.
* Known allergy or sensitivity to ketorolac, ethylene diamine tetraacetic acid (EDTA).
* Prior nasal-septal injury or surgery.
* History of peptic ulcer, gastro-esophageal reflux, or gastrointestinal bleeding.
* History of advanced renal impairment or a risk for renal failure due to volume depletion.
* Clinically significant (in the Investigator's opinion) laboratory test value outside the normal range.
* Use of either (a.) oxycodone at a dose of 30 mg/day or more or (b.) an equivalent dose of another opioid analgesic for a total of more than half of the days during the preceding month.
* The patient requires regular use (daily use in at least 25 days per month) in the 3 months prior to surgery of NSAID's , COX2 inhibitors, tramadol, or acetaminophen at daily dose of more than 2 g for the management of pain.
* Contraindication to the use of morphine, general anesthetics, bupivacaine, ropivacaine, lidocaine, other local anesthetics, muscle relaxants, hydrocodone, ondansetron, or acetaminophen (e.g., significant history of allergic reactions or intolerance to these or related substances).
* Known bleeding diathesis or other disorder or current use of agents affecting coagulation. Deep venous thrombosis prophylaxis of the surgeon's choice is permitted postoperatively.
* Current use of Central Nervous System (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, or Selective Serotonin Reuptake Inhibitors (SSRIs) for pain. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days. The use of lorazepam and other sleep medications, except those containing analgesic properties, are permitted.
* Current diabetes mellitus and HbA1C > 9.5 or a history of prolonged uncontrolled diabetes.
* Use of an antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days.
* Any medical condition that in the investigator's opinion could adversely impact the patient's participation or safety, conduct of the study, or interfere with the pain assessments, including active infection.
* History of drug, prescription medicine, or alcohol abuse that would interfere with the subject's safety or the assessments of efficacy in this trial, in the judgement of the investigator.
* History of nasal mucosal damage or active seasonal allergies, nasal congestion or upper respiratory tract infection sufficient to interfere with intranasal drug delivery.
* Administration of an investigational product within 3 months prior to the first dose of study drug, or scheduled to receive an investigational product, while participating in the study.
* Use of Toradol (ketorolac tromethamine) in any formulation within the past 30 days prior to study entry and throughout study participation.

Max Age: 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-03; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Cmax | Pre-dose, .25, .5, .75, 1, 2, 4, 6 hrs after the 1st dose then prior to each ensuing dose until morning of post-operative Day 2. After a single dose on morning of post-operative Day 2 PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs
  Blood samples will be collected for PK assessment pre-dose, at .25, .5, .75, 1, 2, and 4 hours after the first dose, at 6 hours immediately before the 2nd dose and before each of the next doses up to the dose to be administered on the morning of post operative Day 2. Blood samples will then be collected for PK assessment at 1, 2, 4, 6, 8, 12, and 24 hours after receiving the morning dose on Day 2.
Ctrough | Pre-dose, .25, .5, .75, 1, 2, 4, 6 hrs after the 1st dose then prior to each ensuing dose until morning of post-operative Day 2. After a single dose on morning of post-operative Day 2 PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs
  Blood samples will be collected for PK assessment pre-dose, at .25, .5, .75, 1, 2, and 4 hours after the first dose, at 6 hours immediately before the 2nd dose and before each of the next doses up to the dose to be administered on the morning of post operative Day 2. Blood samples will then be collected for PK assessment at 1, 2, 4, 6, 8, 12, and 24 hours after receiving the morning dose on Day 2.
tmax | Pre-dose, .25, .5, .75, 1, 2, 4, 6 hrs after the 1st dose then prior to each ensuing dose until morning of post-operative Day 2. After a single dose on morning of post-operative Day 2 PK samples will be collected @ 1, 2, 4, 6, 8, 12, & 24 hrs
  Blood samples will be collected for PK assessment pre-dose, at .25, .5, .75, 1, 2, and 4 hours after the first dose, at 6 hours immediately before the 2nd dose and before each of the next doses up to the dose to be administered on the morning of post operative Day 2. Blood samples will then be collected for PK assessment at 1, 2, 4, 6, 8, 12, and 24 hours after receiving the morning dose on Day 2.

CONTACTS AND LOCATIONS:
Overall Officials: Linda M. Mundy, MD, PhD, Study Director — American Regent, Inc.
Locations (4):
- Poland (4):
  - Instytut "Centrum Zdrowia Matki Polki" (Institute "Mother's Memorial Hospital"), Lodz
  - Klinika Chirurgii i Traumatologii Dzieciecej - Dzieciecy Szpital Kliniczny im. prof. Antoniego Gebali, Lublin
  - Regional Hospital of Ludwika Rydygiera in Torun, Torun
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu - Independent Public Clinical Hospital No. 1 in Wroclaw, Wroclaw

IPD SHARING:
Plan to Share IPD: Undecided